CLINICAL TRIAL: NCT01137305
Title: Do Soft Skills Predict Surgical Performance? Do Soft Skills Predict Surgical Performance? A Prospective Randomized Controlled Single Center Educational Trial Evaluating Predictors of Skill Acquisition in Virtual Reality Laparoscopy
Brief Title: Soft Skills and Surgical Performance
Acronym: SSPSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Katja Maschuw, MD, Department of Visceral-, Thoracic- and Vascular Surgery, Philipps- University Marburg, Baldingerstrasse, 35043 Marburg, Germany
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: Katja Maschuw, MD
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Delivery of Health Care
Keywords: Virtual reality; surgical training; Health Care [N]

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: VR- training — Prospective randomization if 50 subjects to either three months of structured VR- training or no training; basic VR- skills assessment and a serial assessment of defined soft skills: self- efficacy, stress- coping and motivation prior to randomization; basic VR- skills measured within seven modules of the VR- simulator LapSim®: "camera and instrument navigation", "coordination", "grasping", "lifting and grasping", "clip applying" and "diathermy cutting" in different levels of difficulty- medium and hard referring to "time to complete task", "economy of instrument motion" and "tissue damage"; intervention group: sessions of 45 minutes each twice a week for three months; control group: no training
  Other Names: Educational trial within surgical trainees

SUMMARY:
Background and hypothesis:

Virtual reality (VR) training in minimal invasive surgery (MIS) is known to be feasible and beneficial in surgical residency. Research on stress- coping in surgical trainees indicate an additional impact of soft skills on VR- performance. Thus to hypothesize soft skills predicting surgical performance in a VR- setting.

Method:

A prospective randomized controlled single center educational trial was carried out to evaluate the impact of structured VR- training and defined soft skills such as self- efficacy, stress- coping and motivation on VR- performance.

DETAILED DESCRIPTION:
Method:

Eligibility criteria were surgical residency not exceeding the first year of surgical training, a limited experience in MIS and informed consent to the study procedures including an anonymized publication of the study data. Limited experience in MIS was defined as camera navigation in laparoscopic cholecystectomies only.

Fifty residents were enrolled and prospectively randomized to either three months of structured VR- training or no training. Every participant underwent a basic VR- skills assessment and a serial assessment of defined soft skills including self- efficacy, stress- coping and motivation prior to randomization.

Basic VR- skills were measured within seven modules of the VR- simulator LapSim® (Surgical Science, Goteborg, Sweden) including "camera and instrument navigation", "coordination", "grasping", "lifting and grasping", "clip applying" and "diathermy cutting". Each module had to be performed in two levels of difficulty- medium and hard. Means of defined parameters of VR- performance were generated. Defined parameters of VR- performance comprised "time to complete task", "economy of instrument motion" and "tissue damage".

Serial assessment of defined soft skills comprised standardized psychological paper- pencil questionnaires regarding self efficacy (GSE), stress coping (SVF 78) and motivation (QCM).

Participants randomized to the intervention group had to pass sessions of 45 minutes each twice a week for three months. Participants randomized to the control group underwent no training at all.

Three months after randomization, VR- performance was assessed likewise. Outcome measurement of VR- performance defined results derived from the most complex module "diathermy- cutting" as endpoint.

The study was approved by the local ethics committee. Participation of the study was voluntary. Data were blinded to the investigators.

The data were descriptively analysed using SPSS® software version 16.0 (SSPS®, Chicago, Illinois, USA). Spearman regression analysis was performed to correlate means of virtual laparoscopic performance and the results derived from serial psychological testing. The differences between the randomized groups were assessed by means of the non- parametric Mann-Whitney- Test regarding all parameters, laparoscopic performance as well psychological scores. Relation of means was carried out using the two- independent t- Test. The level of statistical significance was set at p < 0.050 (two-tailed).

ELIGIBILITY:
Inclusion Criteria:

* surgical residency not exceeding the first year of surgical training
* limited experience in MIS (camera navigation in laparoscopic cholecystectomies only)
* informed consent to study procedures and publication of anonymized data

Exclusion Criteria:

* surgical residency exceeding the first year of surgical training
* experience in MIS exceeding camera navigation in laparoscopic cholecystectomies
* lack of informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
VR- performance after training | Three months
  Outcome measurement comprised defined parameters of VR- performance including "time to complete task", economy of instrument motion" and "tissue damage" within the most complex module "diathermy cutting" as primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Iyad Hassan, MD, Principal Investigator — Department of Visceral-, Thoracic- and Vascular Surgery, Philipps- University Marburg, Germany